CLINICAL TRIAL: NCT06966882
Title: Research on the Real-World Community Application of Large Language Models
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025KYPJ020
Record Dates: First submitted 2025-04-23; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Ophthalmic Diseases (Specific Types Not Restricted)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negative group: Patients manageable at community level；Individuals without ocular pathology
- Positive group: Patients requiring specialist referral

SUMMARY:
There is an imbalance between the supply and demand of eye care services, especially in local communities and remote areas. To address this, it's important to use new intelligent technologies to expand the reach of eye disease screening and treatment. Large language models (LLMs) are a type of deep learning technology that can learn from large amounts of text and generate human-like language to help with medical tasks such as diagnosing diseases and answering health-related questions. The investigator's team has previously developed a localized LLM capable of answering ophthalmology-related medical questions. Building on this, this study plans to use a screening-based trial design to explore how accurately the LLM can make referral decisions for eye diseases, diagnose conditions, recommend appropriate tests, and receive user feedback in real-world community settings. The goal is to improve the ability to screen for eye diseases in grassroots and regional areas.

ELIGIBILITY:
Inclusion Criteria:

* Participants of any age and gender
* Belonging to one of the following ophthalmic categories: Patients requiring specialist referral；Patients manageable at community level；Individuals without ocular pathology
* Voluntary participation with written informed consent

Exclusion Criteria:

* Investigator-determined clinical contraindications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample or primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Metrics for Evaluating Referral Accuracy of Large Language Models: Sensitivity, Specificity, Accuracy, Positive Predictive Value, Negative Predictive Value. | through study completion, up to 1 year.